CLINICAL TRIAL: NCT03573908
Title: A Phase 3b, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial of Linaclotide 290 μg Administered Orally for 12 Weeks Followed by a 4-week Randomized Withdrawal Period in Patients With Irritable Bowel Syndrome With Constipation
Brief Title: A Trial of Linaclotide 290 μg in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCP-103-312
Record Dates: First submitted 2018-06-18; First posted 2018-06-29 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Linaclotide 290 µg (Experimental): Participants receive linaclotide 290 µg orally once daily for 12 weeks during the Treatment Period. At Week 12 participants are rerandomized to receive either linaclotide 290 µg or placebo for 4 weeks in the Randomized Withdrawal Period.
  Interventions: Drug: Linaclotide; Drug: Placebo
- Placebo (Placebo Comparator): Participants receive placebo to linaclotide orally once daily for 12 weeks during the Treatment Period. At Week 12 participants are switched to receive linaclotide 290 µg for 4 weeks during the Randomized Withdrawal Period.
  Interventions: Drug: Linaclotide; Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide — Oral capsule
  Other Names: Linzess
Drug: Placebo — Matching placebo oral capsule

SUMMARY:
To evaluate the efficacy on abdominal symptoms (abdominal bloating, abdominal discomfort, and abdominal pain) and safety of linaclotide 290 μg administered orally to patients with IBS-C.

DETAILED DESCRIPTION:
This study consists of a 12-week Treatment Period followed by 4-week Randomized Withdrawal (RW) Period.

ELIGIBILITY:
Inclusion Criteria:

* Patient has no clinically significant findings on a physical examination and clinical laboratory tests
* Female patients of childbearing potential must agree to use one of the following methods of birth control:

  1. Hormonal contraception
  2. Double-barrier birth control
  3. Maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy
* Patient meets protocol criteria for diagnosis of IBS-C
* Patient demonstrates continued IBS-C symptoms through Pretreatment Period
* Patient maintains a minimum level of compliance with daily diary

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has symptoms of or been diagnosed with a medical condition that may contribute to abdominal pain
* Patient has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilmin Bartolini, PhD, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (78):
- United States (78):
  - Clinical Research Associates, Huntsville, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research, Inc., Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Diagnamics, Inc., Encinitas, California
  - MD Studies, Inc., Fountain Valley, California
  - Paragon Rx Clinical, Inc. - Garden Grove, Garden Grove, California
  - Grossmont Center For Clinical Research, La Mesa, California
  - Facey Medical Foundation, Mission Hills, California
  - Providence Clinical Research, North Hollywood, California
  - Precision Research Institute, San Diego, California
  - Paragon Rx Clinical, Inc.- Santa Ana, Santa Ana, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - St. Joseph Heritage Healthcare, Yorba Linda, California
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Palmetto Research, LLC, Hialeah, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - The Chappel Group Research, Kissimmee, Florida
  - Jesscan Medical Research, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Ocean Blue Medical Research Center, Inc., Miami Springs, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Research Institute of Central Florida, LLC, Winter Park, Florida
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Alan A. Rosen, MD, PA, Baltimore, Maryland
  - Meritus Center For Clinical Research, Hagerstown, Maryland
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Gastroenterology Associates of West Michigan, Wyoming, Michigan
  - Gastrointestinal Associates PA, Flowood, Mississippi
  - St. Louis Center For Clinical Research, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Healthwise Medical Associates, Brooklyn, New York
  - Long Island Gastrointestinal Research Group, LLP, Great Neck, New York
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Concord, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Peters Medical Research, LLC, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Clinical Trials of America - North Carolina, LLC, Winston-Salem, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Hightop Medical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Remington Davis, Inc., Columbus, Ohio
  - Dayton Gastroenterology, Inc., Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Partners In Clinical Research, Cumberland, Rhode Island
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - ClinSearch, LLC, Chattanooga, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - MW Clinical Research Center, Beaumont, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brenner DM, Lacy BE, Ford AC, Bartolini W, Wu J, Shea EP, Bochenek W, Boinpally R, Almansa C. Linaclotide Reduced Response Time for Irritable Bowel Syndrome With Constipation Symptoms: Analysis of 4 Randomized Controlled Trials. Am J Gastroenterol. 2023 May 1;118(5):872-879. doi: 10.14309/ajg.0000000000002064. Epub 2022 Oct 12. PMID 36227782
- [Derived] Chang L, Lacy BE, Moshiree B, Kassebaum A, Abel JL, Hanlon J, Bartolini W, Boinpally R, Bochenek W, Fox SM, Mallick M, Tripp K, Omniewski N, Shea E, Borgstein N. Efficacy of Linaclotide in Reducing Abdominal Symptoms of Bloating, Discomfort, and Pain: A Phase 3B Trial Using a Novel Abdominal Scoring System. Am J Gastroenterol. 2021 Sep 1;116(9):1929-1937. doi: 10.14309/ajg.0000000000001334. PMID 34465695

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment Period (TP, 12 weeks): Participants were randomized 1:1 to linaclotide 290 μg or placebo once daily.
  Randomized Withdrawal Period (4 weeks):
  * Participants randomized to linaclotide 290 μg during TP were rerandomized 1:1 to linaclotide 290 μg or placebo
  * Participants randomized to placebo during TP were allocated to linaclotide 290 μg.
Groups:
- Placebo: Participants were randomized to receive placebo to linaclotide orally once daily for 12 weeks during the Treatment Period.
- Linaclotide 290 µg: Participants were randomized to receive linaclotide 290 µg orally once daily for 12 weeks during the Treatment Period.
- Placebo -> Linaclotide 290 µg: Participants who received placebo orally once daily for 12 weeks during the Treatment Period were switched to receive linaclotide 290 µg for 4 weeks during the Randomized Withdrawal Period.
- Linaclotide 290 µg -> Placebo: Participants who received linaclotide 290 µg orally once daily for 12 weeks during the Treatment Period were rerandomized to receive placebo for 4 weeks in the Randomized Withdrawal Period.
- Linaclotide 290 µg -> Linaclotide 290 µg: Participants who received linaclotide 290 µg orally once daily for 12 weeks during the Treatment Period were rerandomized to continue linaclotide 290 µg for 4 weeks in the Randomized Withdrawal Period.
Period: Treatment Period
Arm/Group | Placebo | Linaclotide 290 µg | Placebo -> Linaclotide 290 µg | Linaclotide 290 µg -> Placebo | Linaclotide 290 µg -> Linaclotide 290 µg
Started | 308 | 306 | 0 | 0 | 0
Completed (Completed 12-week Treatment Period) | 284 | 280 | 0 | 0 | 0
Not Completed | 24 | 26 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 9 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 6 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Other, Not Specified | 4 | 6 | 0 | 0 | 0
Period: Randomized Withdrawal Period
Arm/Group | Placebo | Linaclotide 290 µg | Placebo -> Linaclotide 290 µg | Linaclotide 290 µg -> Placebo | Linaclotide 290 µg -> Linaclotide 290 µg
Started | 0 | 0 | 280 | 138 | 139
Completed | 0 | 0 | 272 | 136 | 137
Not Completed | 0 | 0 | 8 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Other, Not Specified | 0 | 0 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to receive placebo to linaclotide orally once daily for 12 weeks during the Treatment Period.
- Linaclotide 290 µg: Participants randomized to receive linaclotide 290 µg orally once daily for 12 weeks during the Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Linaclotide 290 µg | Total
Number analyzed (Participants) | 308 | 306 | 614
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (14.2) | 46.5 (14.6) | 46.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 241 | 496
  Male | 53 | 65 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 87 | 168
  Not Hispanic or Latino | 227 | 219 | 446
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 198 | 189 | 387
  Black or African American | 70 | 76 | 146
  Asian | 35 | 36 | 71
  Other, Not Specified | 5 | 5 | 10
Abdominal Score (Abdominal Bloating, Abdominal Discomfort, and Abdominal Pain) [Mean (Standard Deviation); unit: score on a scale] — A participant's daily abdominal score was calculated as the average of daily electronic diary (e-diary) abdominal pain, abdominal bloating and abdominal discomfort scores, each based on an 11-point scale of 0 (none) and 10 (very severe). Baseline abdominal score was derived from the eDiary data collected daily in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization.
  score on a scale | 6.46 (1.60) | 6.39 (1.63) | 6.42 (1.61)

OUTCOME MEASURES:

1. Primary Outcome: Overall Change From Baseline in Abdominal Score (Abdominal Bloating, Abdominal Discomfort, and Abdominal Pain) Throughout the Treatment Period
Description: A participant's daily abdominal score was calculated as the average of daily e-diary abdominal pain, abdominal bloating and abdominal discomfort scores, each based on an 11-point scale of 0 (none) and 10 (worst possible). Baseline abdominal score was derived from the eDiary data collected daily in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization. The participant's abdominal score was averaged on a weekly basis, and each weekly change from baseline was calculated for the treatment period and used as the dependent variable in the mixed model with repeated measures (MMRM) model. MMRM results are based on a model with treatment, analysis week, region and treatment-by-week interaction as fixed effects and baseline as a covariate. An unstructured covariance structure was used to model intra-subject correlation with subjects as a random effect.
Time Frame: Baseline (14 days before randomization up to the time of randomization), Treatment Period (Weeks 1-12)
Population: Intent to Treat Population: all randomized participants. Two participants were excluded from the analysis due to missing scores.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Linaclotide 290 µg
Number analyzed (Participants) | 306 | 306
score on a scale | -1.182 (0.109) | -1.898 (0.111)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 290 µg; The overall family-wise Type I error rate for the primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM; Least squares (LS) mean difference = -0.715, 95% CI 2-sided [-0.998 to -0.433] — Least squares (LS) mean difference (linaclotide - placebo)

2. Secondary Outcome: Cumulative Distribution of Change From Baseline in 12-Week Abdominal Score
Description: A participant's daily abdominal score was calculated as the average of daily e-diary abdominal pain, abdominal bloating and abdominal discomfort scores, each based on an 11-point scale of 0 (none) and 10 (worst possible). Baseline abdominal score was derived from the eDiary data collected daily in the Pretreatment Period, specifically the period of time from 14 days before randomization up to the time of randomization. The 12-week abdominal score was the average of the non-missing abdominal scores reported over the course of the treatment period. Change from baseline (BL) was calculated as the 12-week score minus the baseline score. The table presents the percentage of participants whose 12-week change from baseline was less than or equal to the threshold value of the score change (cumulative distribution of change).
Time Frame: Baseline (14 days before randomization up to the time of randomization), Treatment Period (Weeks 1-12)
Population: Intent to Treat Population: all randomized participants. Participants with available 12-week abdominal score.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Linaclotide 290 µg
Number analyzed (Participants) | 306 | 306
percentage of participants
  Change from BL threshold: -9.0 | 0.0 | 0.3
  Change from BL threshold: -8.0 | 0.0 | 0.7
  Change from BL threshold: -7.0 | 0.3 | 1.3
  Change from BL threshold: -6.0 | 0.3 | 2.3
  Change from BL threshold: -5.0 | 2.3 | 6.2
  Change from BL threshold: -4.0 | 4.9 | 14.4
  Change from BL threshold: -3.0 | 11.4 | 24.5
  Change from BL threshold: -2.0 | 23.9 | 40.2
  Change from BL threshold: -1.0 | 42.8 | 58.8
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 290 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon Rank Sum Test; P-value comparing change from baseline distributions by treatment using the Wilcoxon rank sum test 2-sided; Hodges-Lehman Estimated Median Threshold = -0.6, 95% CI 2-sided [-0.88 to -0.35] — 95% confidence interval (CI) for Hodges-Lehmann estimated median threshold was generated by Moses confidence limits method

3. Secondary Outcome: Percentage of 6/12 Week Abdominal Score Responders (Responder Rate)
Description: A 6/12 week abdominal score responder is a participant who meets the weekly abdominal score responder criteria for at least 6 out of the 12 weeks of the Treatment Period. For each week in the Treatment Period, a weekly abdominal score responder is a participant who has an improvement from baseline of at least 2 points (ie, a -2 point change from baseline) in the respective weekly abdominal score. If a participant did not have at least 4 completed eDiary entries for a particular Treatment Period week, the participant was not considered a responder for that week.
  A participant's daily abdominal score was calculated as the average of daily e-diary abdominal pain, abdominal bloating and abdominal discomfort scores, each based on an 11-point scale of 0 (none) and 10 (worst possible). The participant's abdominal score was averaged on a weekly basis, and each weekly change from baseline was calculated for the treatment period.
Time Frame: Baseline (14 days before randomization up to the time of randomization), Treatment Period (Weeks 1-12)
Population: Intent to Treat Population: all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Linaclotide 290 µg
Number analyzed (Participants) | 308 | 306
percentage of participants | 23.4 [18.8 to 28.5] | 40.5 [35.0 to 46.3]
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 290 µg; Test type: Superiority; Difference in Responder Rate = 17.1, 95% CI 2-sided [9.9 to 24.4] — 95% confidence intervals for difference in responder rate are obtained using the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Odds ratio, 95% CI for the Odds Ratio and p-value vs. placebo are obtained from the Cochran-Mantel-Haenszel (CMH) tests controlling for geographic region; Odds Ratio (OR) = 2.20, 95% CI 2-sided [1.55 to 3.12]

4. Secondary Outcome: Overall Change From Baseline in Abdominal Score (Abdominal Bloating, Abdominal Discomfort, and Abdominal Pain) Over Time in the Treatment Period
Description: as for outcome 1
Time Frame: Baseline (14 days before randomization up to the time of randomization), Weeks 1-12
Population: Intent to Treat Population: all randomized participants. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Linaclotide 290 µg
Number analyzed (Participants) | 308 | 306
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 306 | 306
  Change from Baseline at Week 1 | -0.490 (0.085) | -0.925 (0.087)
  Change from Baseline at Week 2: number analyzed (Participants) | 303 | 304
  Change from Baseline at Week 2 | -0.795 (0.102) | -1.423 (0.104)
  Change from Baseline at Week 3: number analyzed (Participants) | 302 | 298
  Change from Baseline at Week 3 | -0.908 (0.110) | -1.592 (0.112)
  Change from Baseline at Week 4: number analyzed (Participants) | 300 | 296
  Change from Baseline at Week 4 | -1.048 (0.115) | -1.731 (0.117)
  Change from Baseline at Week 5: number analyzed (Participants) | 299 | 294
  Change from Baseline at Week 5 | -1.123 (0.118) | -1.891 (0.120)
  Change from Baseline at Week 6: number analyzed (Participants) | 295 | 290
  Change from Baseline at Week 6 | -1.183 (0.122) | -2.014 (0.124)
  Change from Baseline at Week 7: number analyzed (Participants) | 290 | 290
  Change from Baseline at Week 7 | -1.315 (0.125) | -2.073 (0.126)
  Change from Baseline at Week 8: number analyzed (Participants) | 290 | 289
  Change from Baseline at Week 8 | -1.446 (0.130) | -2.110 (0.131)
  Change from Baseline at Week 9: number analyzed (Participants) | 291 | 290
  Change from Baseline at Week 9 | -1.478 (0.129) | -2.181 (0.130)
  Change from Baseline at Week 10: number analyzed (Participants) | 290 | 288
  Change from Baseline at Week 10 | -1.478 (0.130) | -2.197 (0.132)
  Change from Baseline at Week 11: number analyzed (Participants) | 290 | 283
  Change from Baseline at Week 11 | -1.444 (0.131) | -2.288 (0.132)
  Change from Baseline at Week 12: number analyzed (Participants) | 286 | 280
  Change from Baseline at Week 12 | -1.480 (0.133) | -2.347 (0.135)
Statistical Analysis 1: Comparison: Placebo vs Linaclotide 290 µg; Week 12. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM — LS mean difference and p-value were obtained based on an MMRM with treatment, analysis week, geographic region, and treatment-by-week interactions as fixed effects, and baseline score as a covariate; LS mean difference = -0.867, 95% CI 2-sided [-1.219 to -0.515]
Statistical Analysis 2: Comparison: Placebo vs Linaclotide 290 µg; Week 10. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.719, 95% CI 2-sided [-1.062 to -0.376]
Statistical Analysis 3: Comparison: Placebo vs Linaclotide 290 µg; Week 8. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.665, 95% CI 2-sided [-1.007 to -0.322]
Statistical Analysis 4: Comparison: Placebo vs Linaclotide 290 µg; Week 6. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.831, 95% CI 2-sided [-1.151 to -0.511]
Statistical Analysis 5: Comparison: Placebo vs Linaclotide 290 µg; Week 4. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.683, 95% CI 2-sided [-0.982 to -0.383]
Statistical Analysis 6: Comparison: Placebo vs Linaclotide 290 µg; Week 2. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.628, 95% CI 2-sided [-0.888 to -0.368]
Statistical Analysis 7: Comparison: Placebo vs Linaclotide 290 µg; Week 1. The overall family-wise Type I error rate for primary and secondary outcome measures were controlled at the α=0.05 level by employing a fixed-sequence testing procedure. Outcome measures were tested using 10 hypotheses, each comparing linaclotide versus placebo, in the sequence of presentation of statistical analyses in this record. If the hypothesis comparing the 2 groups was statistically significant (α=0.05), then the next hypothesis was to be tested; otherwise, testing would stop; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.435, 95% CI 2-sided [-0.641 to -0.228]
Statistical Analysis 8: Comparison: Placebo vs Linaclotide 290 µg; Week 3. Not part of the fixed-sequence testing procedure; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.683, 95% CI 2-sided [-0.969 to -0.398]
Statistical Analysis 9: Comparison: Placebo vs Linaclotide 290 µg; Week 5. Not part of the fixed-sequence testing procedure; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.768, 95% CI 2-sided [-1.076 to -0.460]
Statistical Analysis 10: Comparison: Placebo vs Linaclotide 290 µg; Week 7. Not part of the fixed-sequence testing procedure; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.758, 95% CI 2-sided [-1.086 to -0.431]
Statistical Analysis 11: Comparison: Placebo vs Linaclotide 290 µg; Week 9. Not part of the fixed-sequence testing procedure; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.703, 95% CI 2-sided [-1.043 to -0.363]
Statistical Analysis 12: Comparison: Placebo vs Linaclotide 290 µg; Week 11. Not part of the fixed-sequence testing procedure; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS mean difference = -0.844, 95% CI 2-sided [-1.189 to -0.498]

ADVERSE EVENTS:
Time Frame: Treatment Period: from first dose of study drug during the Treatment Period to the earlier of: the day after last dose of the Treatment Period and the Day before the first dose of the Randomized Withdrawal (RW) Period. Median duration of treatment was 85 days for both arms during this period. RW Period: from first dose of study drug during the RW Period until the day after the date of the last dose of RW treatment. Median duration of treatment was 29 days for all 3 arms during this period.
Description: Participants in the RW Population (ie, re-randomized or allocated to study drug for the RW Period) who received at least 1 dose of RW treatment were included in the RW Safety Population.
Arm/Group | Placebo | Linaclotide 290 µg | Linaclotide 290 µg -> Linaclotide 290 µg | Linaclotide 290 µg -> Placebo | Placebo -> Linaclotide 290 µg
All-Cause Mortality (participants affected / at risk) | 0/308 | 0/306 | 0/138 | 0/137 | 0/279
Serious Adverse Events (participants affected / at risk) | 2/308 | 4/306 | 1/138 | 0/137 | 1/279
Other Adverse Events (participants affected / at risk) | 15/308 | 26/306 | 5/138 | 4/137 | 21/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=308) | Linaclotide 290 µg (N=306) | Linaclotide 290 µg -> Linaclotide 290 µg (N=138) | Linaclotide 290 µg -> Placebo (N=137) | Placebo -> Linaclotide 290 µg (N=279)
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=308) | Linaclotide 290 µg (N=306) | Linaclotide 290 µg -> Linaclotide 290 µg (N=138) | Linaclotide 290 µg -> Placebo (N=137) | Placebo -> Linaclotide 290 µg (N=279)
Diarrhoea (Gastrointestinal disorders) | 5 | 14 | 3 | 2 | 16
Nasopharyngitis (Infections and infestations) | 9 | 5 | 2 | 2 | 4
Headache (Nervous system disorders) | 3 | 8 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03573908/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03573908/SAP_001.pdf